CLINICAL TRIAL: NCT04116203
Title: Dietary Fish Oil Intervention in Polycystic Ovary Syndrome
Brief Title: Dietary Fish Oil Intervention in Polycystic Ovary Syndrome (PCOS)
Acronym: PCOS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Women and Children's Health Research Institute, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Diabetes Institute (Other); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO00059201
Record Dates: First submitted 2018-05-05; First posted 2019-10-04 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Polycystic Ovary Syndrome; Lipid Metabolism Disorders
Keywords: Polycystic Ovary Syndrome; metabolic and cardiovascular diseases; diabetes; obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Lipid Metabolism Disorders; Cardiovascular Diseases; Diabetes Mellitus; Obesity | interventions — Metformin; Fish Oils; Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: Outcomes at 6 and 12 weeks will be compared to baseline values to determine the efficacy of interventions. Participants will act as their own control in each intervention
Masking Description: This is a randomized open-label parallel study in overweight/obese young women with PCOS, in which the participant will be randomly assigned to one of three treatment arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fish Oil (Other): Fish oil capsules 1200mg 6 tablets/day 12 weeks
  Interventions: Dietary Supplement: Fish Oil
- Metformin (Other): Metformin tablets (500 mg) 2/day 12 weeks
  Interventions: Drug: Metformin
- Fish Oil and Metformin (Other): Combo of other 2 arms
  Interventions: Combination Product: Fish Oil and Metformin

INTERVENTIONS:
Drug: Metformin — Manufacturer's standard 500 mg. Submission Control No.:128147
  Other Names: Metformin Hydrochloride Oral Antihyperglycemic Agent.
  Arms: Metformin
Combination Product: Fish Oil and Metformin — Combo of 2 other arms
  Arms: Fish Oil and Metformin
Dietary Supplement: Fish Oil — NPN: 80028808 Licence Holder: WN Pharmaceuticals Ltd Dosage Form: Capsule, soft Recommended Route of Administration: Oral
  Other Names: Fish Oil; Fish Oil 1200 Mg; Omega-3
  Arms: Fish Oil

SUMMARY:
The primary objective in this proposed study is to determine the effect of dietary fish oil supplementation compared to standard care metformin treatment, and fish oil in combination with metformin on plasma lipids and apoB-remnant lipoprotein metabolism in overweight-obese young women with PCOS.

DETAILED DESCRIPTION:
Specific Objectives;

1. To determine the effect of dietary fish oil supplementation, metformin, and fish oil in combination with metformin on fasting and non-fasting plasma TG, apoB48 and apoB100-lipoprotein concentrations.
2. To determine the physiological mechanisms associated with the effect of dietary fish oil supplementation and metformin on in vivo plasma lipid and apoB-lipoprotein kinetics. We will quantitate the in vivo production and kinetics of plasma TG, apoB48 and apoB100-lipoproteins in plasma and isolated lipoprotein fractions, using established methods.
3. To explore the effects of dietary fish oil supplementation, metformin and fish oil in combination with metformin, on plasma insulin and testosterone, and the association with changes in plasma lipids and apoB-lipoprotein metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age at time of enrollment > 18 to <30 years
* Diagnosis of PCOS: clinical and/or biochemical hyperandrogenemia and menstrual dysfunction and the exclusion of other disorders.
* Overweight-obese (BMI >25 kg/m2) high-risk metabolically-resistant young women.
* Elevated fasting plasma TG (>150 mg/dL) and apoB48-remnant cholesterol lipoproteins (>20 ug/ml).
* Impaired insulin sensitivity (glucose 100-125 mg/dL and/or insulin >15 (uM/ml); and
* May be diagnosed with T2D (blood glucose >126 mg/dL).

Exclusion Criteria:

* Pregnancy
* Lactating women
* Recent illness that the investigator determines to pose a potential risk for the participant
* Concomitant medications that influence metabolism (e.g. statins)
* Excessive alcohol consumption, as determined by the investigator.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The focus of this study is on overweight-obese high-risk metabolically-resistant young women (aged 18-30 yrs) newly diagnosed with PCOS
Enrollment: 52 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Plasma Triglycerides and apoB-lipoprotein remnants in non-fasting and fasted state | At baseline and postintervention at 12 weeks
  reported as mean +/- SEM

SECONDARY OUTCOMES:
Plasma insulin and glucose | At baseline and postintervention at 12 weeks
  reported as mean +/- SEM
Plasma hormones, testosterone, SHBG, Estrogen | At baseline and postintervention at 12 weeks
  reported as mean +/- SEM

CONTACTS AND LOCATIONS:
Overall Officials: Donna F Vine, PhD, Principal Investigator — Associate Professor
Locations (2):
- Canada (2):
  - 9-111 Endocrinology Department, UofA Hospital, Edmonton, Alberta
  - 2-004 Li Ka Shing Centre, UofA, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No
There will be no sharing with other researchers.

REFERENCES:
- [Result] Vine DF, Wang Y, Jetha MM, Ball GD, Proctor SD. Impaired ApoB-Lipoprotein and Triglyceride Metabolism in Obese Adolescents With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2017 Mar 1;102(3):970-982. doi: 10.1210/jc.2016-2854. PMID 27997268